CLINICAL TRIAL: NCT04504448
Title: A Randomized, Double-blind, Placebo-controlled, Sequential Parallel Group, Single Ascending Doses (SAD) Study Following Oral Administration in Healthy Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Food Effect of HNC664
Brief Title: A Study of HNC664 in Healthy Subjects to Evaluate the Safety, Tolerability, and Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Henovcom Bioscience Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HNC664-101
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- HNC664 capsules (Experimental): HNC664 capsules,single ascending doses Single dose
  Interventions: Drug: HNC664 capsules Single dose
- HNC664 placebos (Placebo Comparator): HNC664 placebos,single ascending doses Single dose
  Interventions: Drug: HNC664 placebos Single dose
- HNC664 capsules FED (Experimental): HNC664 capsules,food effect,Single dose
  Interventions: Drug: HNC664 capsules FED

INTERVENTIONS:
Drug: HNC664 capsules Single dose — HNC664 capsules,single ascending doses Single dose, PO,starting dose of 40mg escalating up to 500mg
  Other Names: HNC664 capsules
  Arms: HNC664 capsules
Drug: HNC664 placebos Single dose — HNC664 placebos single ascending doses,PO,Single dose, matching placebo
  Other Names: HNC664 placebos
  Arms: HNC664 placebos
Drug: HNC664 capsules FED — HNC664 capsules,single doses Single dose, PO,food effect（dosage will be based on data from SAD cohorts and decided by the IDRC）
  Other Names: HNC664 capsules
  Arms: HNC664 capsules FED

SUMMARY:
The purpose of this First-in-Human study is to evaluate the safety , tolerability，PK and PD after single ascending of HNC664 given to healthy subjects, compared to placebo. Also, food effect will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer, age 18-65 years
* BMI between 18-32 kg/m2,and body weight not less than 50.0kg.

Exclusion Criteria:

* Any condition that might interfere with the procedures or tests in this study
* Drug or alcohol abuse
* Smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events and concomitant medications | Between screening and 7-9 days after the last dose
  To evaluate the safety and tolerability of HNC664 in comparison with placebo after a single oral dose in healthy subjects in terms of AEs and CMs.
Number of subjects with vital sign measurements | Between screening and 7-9 days after the last dose
  To evaluate the safety and tolerability of HNC664 in comparison with placebo after a single oral dose in healthy subjects in terms of abnormal vital signs
Number of subjects with clinical laboratory test results | Between screening and 7-9 days after the last dose
  To evaluate the safety and tolerability of HNC664 in comparison with placebo after a single oral dose in healthy subjects in terms of abnormal clinical laboratory test results
Number of subjects with 12-lead ECGs | Between screening and 7-9 days after the last dose
  To evaluate the safety and tolerability of HNC664 in comparison with placebo after a single oral dose in healthy subjects in terms of abnormal 12-lead ECGs
Number of subjects with physical examinations | Between screening and 7-9 days after the last dose
  To evaluate the safety and tolerability of HNC664 in comparison with placebo after a single oral dose in healthy subjects in terms of abnormal physical examinations

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron, Baltimore, Maryland, United States